CLINICAL TRIAL: NCT03290729
Title: Wedge Implant for Minimally Invasive Treatment of Narrow Crests: a Prospective Multi-center Clinical Study
Brief Title: Wedge Implant Narrow Crests: Multi-center Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Piezosurgery Academy (Other)
Responsible Party: Principal Investigator, Mr. Claudio Stacchi, DDS, MSc, President of the Academy, International Piezosurgery Academy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REX_i
Record Dates: First submitted 2017-07-21; First posted 2017-09-25 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Alveolar Bone Loss
Keywords: wedge implants; atrophic bone
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: multicenter single cohort prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- narrow ridge (Experimental): edentulous site with crestal bone width comprised between 3,5 and 5 millimeters wedge shape implants insertion
  Interventions: Procedure: wedge shape implants insertion

INTERVENTIONS:
Procedure: wedge shape implants insertion — Narrow dental implants inserted in narrow ridges

SUMMARY:
This study was designed as a multicentric prospective clinical trial to assess the clinical, biological and patient's perceived success of new wedge-shaped dental implants inserted in narrow ridges.

DETAILED DESCRIPTION:
Due to the loss of dental elements, the bone crest undergoes a significant remodeling. Bone resorption begins immediately after dental extraction with a 40-60% reduction in horizontal and vertical direction of the alveolar ridge during the first 2 years. The most significant bone loss after tooth extraction occurs within the first 3 months, although modeling and remodeling of the alveoli have a great variability of time: bone structure and organization may not be complete even 24 weeks after dental extraction.

It is now known that crestal remodeling is closely related to the disappearance of the bundle bone, which is more representative of the buccal appearance of the alveolus. Its disappearance, especially in thin periodontal biotopes, can lead to significant recessions of hard and soft tissues.

Moreover, with a variable percentage, in many patients, crestal resorption continues over time due to a combination of factors involved: anatomical, metabolic and mechanical. Among these, the use of removable total or partial dentures can play an important role in accelerating the resurfacing process.

With these premises, it is common to find patients with atrophic crests when processing plans that provide implant support prosthetic rehabilitation.

A crestal bone thickness of at least 6 mm in the buco-lingual sense is considered sufficient to safely place a plant with a diameter of 4 mm. But when the width is lower, a variety of procedures and techniques have been proposed in literature that allow recreate the volumes needed for implant placement.

Horizontal lifting techniques with bone blocks (autologous, alloplastic, xeno-graft), guided bone regeneration, crest expansion technique have demonstrated a good long-term predictability of the inserted devices. However, some negatives related to these techniques need to be considered, such as increased morbidity for the patient, demand for advanced surgical skills for the operator, increased treatment costs, and increased therapy times.

Because of these observations, a new implant design has been proposed for specific use in narrow ridges. Its wedge shape and press-fit insertion make it possible to position it with a minimally invasive preparation of the implant site, performed with ultrasound technique.

Therefore, the use of this implant could allow effective and minimally invasive treatment of narrow edentulous crests up to 4 mm, with significant benefits to the patient in terms of morbidity, treatment costs and time.

Twelve clinical centers will treat patients with insertion of wedge-shaped implants in thin crests with a specific surgical protocol and clinical outcomes will be collected and analyzed.

The chosen medical device will be the Rex Tissue Level implant System. For each implant inserted, the clinical parameters will be recorded up to 5 years after insertion.

In addition, intermediate evaluations will be carried out at 1 year and 3 years after installation.

ELIGIBILITY:
Inclusion Criteria:

1. indications for prosthetic rehabilitation supported by implants in the upper or lower arch, based on accurate diagnosis and treatment planning;
2. the bone crest must be completely healed (at least six months after the tooth loss);
3. residual bone ridge width between 3.5 and 5 mm, at least 3 mm in apical direction;
4. presence of at least 10 mm bone height available for implant placement;
5. age of the patient> 18 years;
6. The patient must not carry any removable prosthesis on the treated area;
7. the patient must be able to follow the protocol of study;
8. informed written consent

Exclusion Criteria:

1. acute myocardial infarction over the last 2 months;
2. uncontrolled coagulation disorders;
3. unmanaged diabetes (HBA1c> 7.5);
4. radiotherapy to the head area in the last 24 months;
5. immunocompromised, HIV positive or chemotherapy patients over the past 5 years;
6. present or past treatment with intravenous bisphosphonates;
7. psychological or psychiatric problems;
8. abuse of alcohol or drugs;
9. uncontrolled periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
implant survival rate | 1 year after surgery
  health of the inserted implants

SECONDARY OUTCOMES:
surgical procedure evaluation | during surgery
  handling assessment of the implant system by the surgeons
surgical procedure evaluation | 1 hour after surgery
  assessment of the invasivity of the surgical procedure from the patient
implant stability 14 | 14 days after surgery
  resonance frequence analysis of the implant
implant stability 1 month | 1 month after surgery
  resonance frequence analysis of the implant
implant stability 2 months | 2 months after surgery
  resonance frequence analysis of the implant
implant stability 3 months | 3 months after surgery
  resonance frequence analysis of the implant
implant stability 4 months | 4 months after surgery
  resonance frequence analysis of the implant
implant stability 5 months | 5 months after surgery
  resonance frequence analysis of the implant
implant stability 6 months | 6 months after surgery
  resonance frequence analysis of the implant
implant stability 1 year | 1 year after surgery
  resonance frequence analysis of the implant
implant stability 3 years | 3 years after surgery
  resonance frequence analysis of the implant
implant stability 5 years | 5 years after surgery
  resonance frequence analysis of the implant

CONTACTS AND LOCATIONS:
Overall Officials: claudio stacchi, Dr., Principal Investigator — Piezosurgery Academy
Locations (1):
- Piezosurgery Academy, Parma, PR, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiapasco M, Zaniboni M. Clinical outcomes of GBR procedures to correct peri-implant dehiscences and fenestrations: a systematic review. Clin Oral Implants Res. 2009 Sep;20 Suppl 4:113-23. doi: 10.1111/j.1600-0501.2009.01781.x. PMID 19663958
- [Background] Danza M, Guidi R, Carinci F. Comparison between implants inserted into piezo split and unsplit alveolar crests. J Oral Maxillofac Surg. 2009 Nov;67(11):2460-5. doi: 10.1016/j.joms.2009.04.041. PMID 19837318
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475